CLINICAL TRIAL: NCT04734457
Title: Final Height in Patients With Congenital Hypothyroidism Diagnosed by Neonatal Screening
Brief Title: Final Height in Patients With CH Diagnosed by the Screening
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mohamed Nader, Principal Investigator, Ain Shams University
Other Study IDs: Final height in CH patients
Record Dates: First submitted 2021-01-11; First posted 2021-02-02 (Actual); Last update posted 2021-10-05 (Actual); Status verified 2021-10

CONDITIONS: Congenital Hypothyroidism
Keywords: Final Height; Neonatal screening
MeSH Terms: conditions — Congenital Hypothyroidism | interventions — Thyroxine; Neonatal Screening

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Levothyroxin — We assess the effect of early diagnosis of CH by neonatal screening and start of treatment on the final height of the patients
  Other Names: neonatal screening

SUMMARY:
The aim of this study is to evaluate longitudinal growth and final height in patients with Congenital Hypothyroidism detected by neonatal screening and factors affecting it.

DETAILED DESCRIPTION:
Linear growth and final height are reported as rather normal in patients with CH diagnosed through the screening and the target height is the most important factor determining linear growth. Data on final height in patients with CH suggest that adult height is significantly correlated with parental height and the mean L-Thyroxine daily dose administered over the first 6 months of treatment. The lowest recommended dose during this period is 8.5μg/kg/day. Periodical adjustments of L-Thyroxine daily dose should be guided by clinical observation and serum free T4 levels.

To our knowledge this is the first study from our center to assess final height in patients with congenital hypothyroidism diagnosed through the Egyptian neonatal screening program.

A complex network of endocrine signals stimulates the process of longitudinal growth including growth hormone, insulin-like growth factor-1, glucocorticoids, thyroid hormone, estrogen, androgens, vitamin D and leptin.

Thyroid hormones are essential for development and normal bone growth. Biochemical studies have shown that thyroid hormones can affect the expression of various bone markers in the serum, reflecting changes in bone remodeling which involves both osteoblastic and osteoclastic activities.

Thyroid hormones act through chondrocytes bearing thyroid hormone receptors (TRs) to modulate growth plate proliferation, differentiation and vascular invasion. Several mechanisms mediate these functions including direct action on the chondrocytes, osteoblasts and mast cells. It also works through interaction with other hormones and growth factors acting in endocrine, paracrine and autocrine fashions.

Overall, T3 acts via TRα in chondrocytes and osteoblasts to regulate intramembranous and endochondral ossification and control the rate of linear growth, bone maturation and mineralization,T4 induces the expression of both type II and X collagen and chondrocyte hypertrophy.

Hypothyroidism in children causes growth arrest, delayed bone maturation, and epiphyseal dysgenesis that can result in short stature and delayed closure of the epiphyses.

In severe undiagnosed cases, complete post-natal growth arrest and skeletal dysplasia occurs with characteristic X-ray features including stippled epiphyses reflecting epiphyseal dysgenesis, congenital hip dislocation, vertebral immaturity, scoliosis, patent fontanelles and sutures and delayed eruption of teeth.

Prompt treatment of patients suffering from CH with thyroid hormone replacement induces a period of rapid catch-up growth in which skeletal maturation and bone age are also accelerated. Ultimately, normal adult height can be expected.

It is controversial whether factors as the degree of hypothyroidism at diagnosis, the timing of the onset of treatment and the doses of replacement L-thyroxine (L-T4) affect linear growth in children with congenital hypothyroidism, detected by screening and treated from early infancy

ELIGIBILITY:
Inclusion Criteria:

* Patients having a documented history of CH diagnosed by Egyptian neonatal screening program.
* Patients receiving L-thyroxine (L-T4) since the diagnosis is established.

Exclusion Criteria:

* Patients who are non-compliant on L-thyroxine (L-T4) and failed to follow up at the clinic on regular basis.
* Patients who were missed from diagnosis by neonatal screening.
* Patients with associated hormonal disorders affecting same parameters concerned in the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All the patients suffering from CH diagnosed by Egyptian neonatal screening program and have a documented history of CH who received treatment at endocrinology clinic, Children's Hospital, Ain Shams University.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2021-11-02 (Estimated); Primary Completion 2022-03-01 (Estimated); Study Completion 2022-04-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of change of Final Height in patients with Congenital Hypothyroidism diagnosed by neonatal screening | Since the diagnosis is established by neonatal screening during first week of life height will be assessed every 6 months with follow up throughout the study period until the study subject reaches an average of 18 years of age( final height reached).
  The investigators assess the effect of early diagnosis and early levothyroxine start on the change in longitudinal growth in patients with Congenital Hypothyroidism.

CONTACTS AND LOCATIONS:
Overall Officials: Wessam Mouharram, PhD, Study Director — Ain Shams University; Rana Mahmoud, PhD, Study Director — Ain Shams University
Locations (1):
- Ain Shams University, Cairo, Abbasiya, Egypt

REFERENCES:
- [Background] Bain P, Toublanc JE. Adult height in congenital hypothyroidism: prognostic factors and the importance of compliance with treatment. Horm Res. 2002;58(3):136-42. doi: 10.1159/000064489. PMID 12218379
- [Result] Bassett JH, Williams AJ, Murphy E, Boyde A, Howell PG, Swinhoe R, Archanco M, Flamant F, Samarut J, Costagliola S, Vassart G, Weiss RE, Refetoff S, Williams GR. A lack of thyroid hormones rather than excess thyrotropin causes abnormal skeletal development in hypothyroidism. Mol Endocrinol. 2008 Feb;22(2):501-12. doi: 10.1210/me.2007-0221. Epub 2007 Oct 11. PMID 17932107
- [Result] Bauer AJ, Wassner AJ. Thyroid hormone therapy in congenital hypothyroidism and pediatric hypothyroidism. Endocrine. 2019 Oct;66(1):51-62. doi: 10.1007/s12020-019-02024-6. Epub 2019 Jul 26. PMID 31350727
- [Result] Cole TJ, Freeman JV, Preece MA. Body mass index reference curves for the UK, 1990. Arch Dis Child. 1995 Jul;73(1):25-9. doi: 10.1136/adc.73.1.25. PMID 7639544
- [Result] Dickerman Z, De Vries L. Prepubertal and pubertal growth, timing and duration of puberty and attained adult height in patients with congenital hypothyroidism (CH) detected by the neonatal screening programme for CH--a longitudinal study. Clin Endocrinol (Oxf). 1997 Dec;47(6):649-54. doi: 10.1046/j.1365-2265.1997.3181148.x. PMID 9497870
- [Result] Huffmeier U, Tietze HU, Rauch A. Severe skeletal dysplasia caused by undiagnosed hypothyroidism. Eur J Med Genet. 2007 May-Jun;50(3):209-15. doi: 10.1016/j.ejmg.2007.02.002. Epub 2007 Mar 12. PMID 17433800
- [Result] Nilsson O, Marino R, De Luca F, Phillip M, Baron J. Endocrine regulation of the growth plate. Horm Res. 2005;64(4):157-65. doi: 10.1159/000088791. Epub 2005 Oct 4. PMID 16205094
- [Result] Salerno M, Micillo M, Di Maio S, Capalbo D, Ferri P, Lettiero T, Tenore A. Longitudinal growth, sexual maturation and final height in patients with congenital hypothyroidism detected by neonatal screening. Eur J Endocrinol. 2001 Oct;145(4):377-83. doi: 10.1530/eje.0.1450377. PMID 11580992
- [Result] Tanner JM, Goldstein H, Whitehouse RH. Standards for children's height at ages 2-9 years allowing for heights of parents. Arch Dis Child. 1970 Dec;45(244):755-62. doi: 10.1136/adc.45.244.755. PMID 5491878
- [Result] Whitney GA, Kean TJ, Fernandes RJ, Waldman S, Tse MY, Pang SC, Mansour JM, Dennis JE. Thyroxine Increases Collagen Type II Expression and Accumulation in Scaffold-Free Tissue-Engineered Articular Cartilage. Tissue Eng Part A. 2018 Mar;24(5-6):369-381. doi: 10.1089/ten.TEA.2016.0533. Epub 2017 Jul 7. PMID 28548569
- [Result] Williams GR. Role of thyroid hormone receptor-alpha1 in endochondral ossification. Endocrinology. 2014 Aug;155(8):2747-50. doi: 10.1210/en.2014-1527. No abstract available. PMID 25036648
- [Result] Williams GR, Bassett JHD. Thyroid diseases and bone health. J Endocrinol Invest. 2018 Jan;41(1):99-109. doi: 10.1007/s40618-017-0753-4. Epub 2017 Aug 29. PMID 28853052